CLINICAL TRIAL: NCT00854061
Title: Study of T-PRED(TM) Compared to Pred Forte(R) II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CL-PKT-0415083-P
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- T-Pred (Experimental): Tobramycin prednisolone acetate combination
  Interventions: Drug: T-Pred
- Pred Forte (Active Comparator): Prednisolone acetate
  Interventions: Drug: Pred Forte

INTERVENTIONS:
Drug: T-Pred — sterile ophthalmic solution
  Arms: T-Pred
Drug: Pred Forte — sterile ophthalmic solution
  Arms: Pred Forte

SUMMARY:
Study of T-PRED(TM) Compared to Pred Forte(R)

DETAILED DESCRIPTION:
This study was a multi-center, randomized, double-masked, bioequivalence study. A total of 172 participants undergoing bilateral cataract surgery were assigned investigational product to each eye according to a computer-generated randomization list for each of 2 study variables: treatment with T-PRED or Pred Forte in the first eye undergoing cataract extraction and the aqueous humor sampling time point.

The investigator determined which eye was clinically suited for the first operative procedure; treatment of this eye was randomized to either T-PRED or Pred Forte. The second eye received the other study treatment (RP if the first eye received T-PRED; T-PRED if the first eye received Pred Forte) at the time of the second cataract extraction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

Exclusion Criteria:

* No active or adverse disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Participants received both treatment groups, one in each eye.
  A total of 172 participants undergoing bilateral cataract surgery were assigned investigational product to each eye according to a computer-generated randomization list for each of 2 study variables: treatment with T-PRED or Pred Forte in the first eye undergoing cataract extraction and the aqueous humor sampling time point.
  The investigator determined which eye was clinically suited for the first operative procedure (surgery); treatment of this eye was randomized to either T-PRED or Pred Forte. The second eye received the other study treatment (RP if the first eye received T-PRED; T-PRED if the first eye received Pred Forte) at the time of the second cataract extraction.
Period: Overall Study
Arm/Group | All Study Participants
Started | 172
Completed 1st Surgery (T-PRED in One Eye and Pred Forte in the Other Eye) | 162
Completed 2nd Surgery (T-PRED and Pred Forte in Opposite Eyes Compared to 1st Surgery) | 149
Completed | 149
Not Completed | 23

BASELINE CHARACTERISTICS:
Groups:
- Overall: Participants received both treatment groups, one in each eye. The treatment assigned to an eye (right or left) was randomly assigned.
Arm/Group | Overall
Number analyzed (Participants) | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: Means Aqueous Humor Prednisolone Acetate Concentration
Time Frame: 35 days
Population: Participants received both treatment groups, one in each eye. The treatment assigned to an eye (right or left) was randomly assigned.
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Arm/Group | T-Pred | Pred Forte
Number analyzed (Participants) | 162 | 162
Number analyzed (eyes) | 81 | 81
ng/mL | 100.02 (9.61) | 131.65 (9.61)

ADVERSE EVENTS:
Time Frame: 35 days
Description: The safety population was comprised of participants who received study treatment and had at least one post-baseline safety assessment. Participants received both treatment groups, one in each eye. The treatment assigned to an eye (right or left) was randomly assigned.g
Arm/Group | T-Pred | Pred-Forte
Serious Adverse Events (participants affected / at risk) | 1/162 | 1/162
Other Adverse Events (participants affected / at risk) | 0/162 | 0/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T-Pred (N=162) | Pred-Forte (N=162)
IOL dislocation (Eye disorders) | 1 | 0
Vitritis (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.